CLINICAL TRIAL: NCT06199635
Title: Evaluate the Initial Safety and Device Functionality of the SFM Anastomosis Device for a Primary Sleeve Gastrectomy Duodenal-Ileal Anastomosis (SNAP-S) or After Primary Sleeve Gastrectomy (SNAP-PS) or to Create a Jejuno-Jejunostomy in a Roux-en-Y Gastric Bypass (J-J)
Brief Title: Early Feasibility for Safety & Device Functionality of SFM Anastomosis Device Used in 3 Procedures (SNAP-S) or (SNAP-PS) or (J-J)
Acronym: GIW-SFM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: GI Windows, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GIW 23-005
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SNAP-S (Experimental): Self-Forming Magnetic (SFM) Anastomosis Device and Delivery System being used to to Create a Primary Sleeve Gastrectomy Duodenal-Ileal Anastomosis
  Interventions: Device: Self-Forming Magnetic Anastomosis Device and Delivery System
- SNAP-PS (Experimental): Self-Forming Magnetic (SFM) Anastomosis Device and Delivery System being used to to Create a Duodenal-ileal Anastomosis years after a Primary Sleeve Gastrectomy)
  Interventions: Device: Self-Forming Magnetic Anastomosis Device and Delivery System
- J-J (Experimental): Self-Forming Magnetic (SFM) Anastomosis Device and Delivery System being used to to Create a Jejuno-Jejunostomy in a Roux-en-Y Gastric Bypass
  Interventions: Device: Self-Forming Magnetic Anastomosis Device and Delivery System

INTERVENTIONS:
Device: Self-Forming Magnetic Anastomosis Device and Delivery System — Self-Forming Magnetic Anastomosis Device to create a gastrointestinal anastomosis

SUMMARY:
The objectives of this study are to assess the initial safety and device functionality of the SFM Anastomosis System including delivery systems when used to create a duodenal-ileal (D-I) anastomosis either during sleeve gastrectomy (i.e., SNAP-S procedure) or patients with prior sleeve gastrectomy who experience inadequate weight loss (i.e., SNAP-PS procedure) or a Roux-en-Y gastric bypass jejuno-jejunostomy. Additionally, the study is designed to evaluate the potential of these procedures to induce weight loss and to improve metabolic comorbidities in obese subjects.

DETAILED DESCRIPTION:
This is a multi-arm, single-center, early feasibility study to evaluate the use of the SFM Anastomosis System for creation of a Duodenal-ileal anastomosis in participants undergoing primary sleeve gastrectomy (SNAP-S cohort) or who have experienced inadequate weight loss following sleeve gastrectomy (SNAP-PS cohort) defined to be failure to achieve a minimum 50% EWL at least 18 months post sleeve gastrectomy or creating the jejuno-jejunostomy anastomosis in a Roux-en-Y gastric bypass. Adult male and female subjects between the ages of 18 and 65 years-old who are candidates for the primary or revisional surgery will be considered for participation.

Patients appearing to meet basic eligibility criteria and who sign the study specific consent form will be screened for enrollment into this study and will be assessed by a multidisciplinary research team with pre-procedure nutritional and medical evaluation (including psychological and behavioral evaluation by an internist/bariatrician).

Subjects meeting the inclusion and exclusion criteria and enrolled into the study will undergo a procedure using the SFM anastomosis device in which the duodenum will be connected to the ileum with the creation of an anastomosis using the SFM device and delivery systems. For subjects undergoing concurrent sleeve gastrectomy and D-I anastomosis (SNAP-S cohort) it is anticipated that the D-I diversion will be created after the sleeve gastrectomy (unless the investigator determines that the reverse order is more appropriate for a particular subject). For subjects undergoing a Roux-en-Y gastric bypass, the standard surgical protocol will be followed at the institution coupled with the minor changes required to connect the SFM device.

ELIGIBILITY:
Inclusion Criteria:

* All Subjects:

  1. Age 18-65 years at screening
  2. For the primary or post sleeve gastrectomy Anastomosis procedures (SNAP-S/SNAP-PS)- Obesity with Body Mass Index (BMI) ≥ 35 kg/m2 but ≤ 55 kg/m2 at time of screening with or without comorbidities at time of screening. If subject has obesity-related comorbidities such as hypertension, dyslipidemia, and sleep apnea, these comorbidities must be well-controlled
  3. For the Roux-en-Y gastric bypass jejuno-jejunostomy procedure (J-J) - Obesity with Body Mass Index (BMI) ≥ 35 kg/m2 but ≤50 kg/m2 with or without comorbidities at time of screening. If subject has obesity-related comorbidities such as hypertension, dyslipidemia, and sleep apnea, these comorbidities must be well-controlled.
  4. Able to understand and sign informed consent document
  5. Patient lives, and intends to remain, within a 150-km radius of study center for 12 months
  6. Willing to commit to sustained healthy behaviors that include diet, eating and exercise habits for the duration of the trial
  7. Willing to refrain from smoking during the study follow-up period
  8. If subject is female, she must commit to not becoming pregnant for 12 months and agree to use of contraceptives during this period and may not be nursing

Exclusion Criteria:

* 1. Known or suspected allergy to nickel, titanium or Nitinol

  2. Type 1 Diabetes

  3. Uncontrolled T2DM Fasting glucose ≥ 200 mg/dl (11.1 mmol/L) and/or hemoglobin A1c >10 or use of injectable insulin

  4. Any documented conditions for which endoscopy and/or laparoscopy would be contraindicated or history of previous technically difficult or failed endoscopy

  5. Contraindication to general anesthesia

  6. Clinically significant finding during procedural endoscopy such as presence of an unhealed ulcers, bleeding lesions, tumors or ischemic or necrotic tissue at target magnet deployment site

  7. Congenital or acquired anomalies of the GI tract, including atresia, stenosis, prior obstruction or malrotation

  8. Presence of a duodenal diverticulum (>10mm)

  9. Any previous major surgery on the stomach, duodenum, hepatobiliary tree (excluding laparoscopically removed gallbladder), pancreas or right colon

  10. History of chronic gastrointestinal disease (e.g., cirrhosis, inflammatory bowel disease) that in the opinion of the Investigator may preclude safe and complete study participation

  11. Uncontrolled severe hypertension (blood pressure >160/100mmHg)

  12. Pre-existing severe comorbid cardio-respiratory disease (e.g., congestive heart failure, uncontrolled cardiac arrhythmia, coronary artery disease, chronic obstructive lung disease requiring supplemental oxygen, pulmonary embolism, Myocardial Infarction with prior 6 months)

  13. Liver biochemistries (ALT and AST) ≥ 3 times the upper limit of normal

  14. Uncorrectable coagulation disorder (platelets < 100,000, PT >2 seconds above upper normal limit or INR >1.5) at time of procedure, Note: management of anti-platelet medications, when applicable, will follow standard practices of the institution

  15. Uncorrectable anemia (Hemoglobin < 11 g/dL in women and <12.5 g/dL in men)

  16. Specific genetic or hormonal cause of obesity such as Prader -Willi syndrome

  17. For females of child-bearing potential: Pregnancy or desire to be pregnant during the study

  18. Concurrent condition anticipated to require MR imaging within the first 2 months after the study procedure

  19. Diagnosed Bulimia Nervosa or Binge Eating Disorder (using DSM-5 criteria)

  20. Physical or mental disability or psychological illness that in the opinion of the Investigator would be a contraindication for bariatric surgery

  21. Subject is immunocompromised (e.g., active treatment for malignancies, hematologic malignancy, on immunosuppressive therapy, moderate or severe primary immunodeficiency, advanced or untreated HIV, active treatment with high-dose corticosteroids (i.e.,20 or more mg of prednisone or equivalent per day when administered for 2 or more weeks prior to surgery) or other immunosuppressive or immunomodulatory agents.

  22. Subject has an active or suspected infection at the surgical site or a CDC Class 3/contaminated or Class 4/dirty-infected surgical wound. Subject is not appropriate for inclusion in the clinical trial, per the medical opinion of the Principal Investigator"

  23. Other prior or concurrent conditions that in the opinion of the Investigator would be unlikely to receive clinical benefit from the study procedure or participation in the study may compromise patient safety or study objectives such as the presence/diagnosis of a severe and evolutive life threatening pathology unrelated to obesity including but not limited to: ongoing infection, chronic pancreatitis, severe hepatic dysfunction, or renal dysfunction (GFR <60mL/min/1.73m2)

  24. Any form of substance abuse or psychiatric disorder that in the opinion of the investigator could interfere with the conduct of the study

  25. (Women only) Pregnancy at screening (+ urine hCG) or unwilling to use contraception throughout study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary Effectiveness Endpoint: | 30 days
  Ability to create the anastomosis with SFM without the need for open conversion or use of additional laparoscopic/endoscopic anastomoses devices (endoscopic/laparoscopic suture devices or staplers - except for closure of the laparoscopic enterotomy).
Primary Safety Endpoint: | 30 days
  The primary safety endpoint for this study is "Freedom from anastomosis adverse events" or "FFAAE" within 30 days including American College of Surgeons (ACS) Grade B/C anastomosis leak (requiring active therapeutic intervention/re-laparotomy), anastomotic bleeding, and small bowel obstruction. All adverse events will be documented.

SECONDARY OUTCOMES:
Total Body Weight Loss (TBWL) | 12 months
  Percent total body weight loss (TBWL) calculated as: % TBWL = [((initial weight - final weight)) ⁄ (initial weight)] × 100
Percent Responders | 12 Months
  Percent of patients losing at least 10% of their baseline weight (i.e., weight at time of study procedure).

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Bhandari, MD, Principal Investigator — Chief of Surgery
Locations (2):
- Clinica Colonial Hospital, Santiago, Huechuraba, Región Metropolitana, Chile
- Bhandari Hospital & Research Centre, Indore, Madhya Pradesh, India

IPD SHARING:
Plan to Share IPD: No